CLINICAL TRIAL: NCT07264920
Title: Pediatric Electrocutaneous Analgesia for Children Experiencing Neuropathic Pain
Acronym: PEACE-NP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00520236
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Neuropathic Pain; Chronic Pain
Keywords: pediatric oncology; chronic pain; neuropathic pain
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment - Scrambler Therapy MC-5A Device (Experimental): Surface electrodes will be placed near the pain site to deliver low-level electrical signals that "scramble" pain messages into non-painful sensations.
  Interventions: Device: Scrambler Therapy MC-5A Device

INTERVENTIONS:
Device: Scrambler Therapy MC-5A Device — Scrambler Therapy is a non-invasive electrocutaneous analgesia technique used to treat neuropathic pain. Each session lasts approximately 30-45 minutes and involves placing surface electrodes near the pain site to deliver low-level electrical signals that "scramble" pain messages into non-painful sensations. Pain intensity will be measured before and after each session.

SUMMARY:
This is a study evaluating the Scrambler Therapy device as a non-invasive treatment for neuropathic pain in pediatric oncology patients with metastatic bone disease. The primary goal is to assess changes in pain intensity and medication use, aiming to improve quality of life and reduce reliance on systemic pain medications.

DETAILED DESCRIPTION:
Eligible participants (ages 5-26) will undergo 5 to 10 therapy sessions over 1-2 weeks, with pain assessed before and after each session using age-appropriate scales. Additional assessments include the PainDETECT questionnaire and follow-ups at 1, 3, and 6 months to evaluate durability of pain relief and changes in medication use.

The study will enroll up to 70 participants over 5 years, with an expected evaluable sample size of 60. Statistical analyses will compare pre- and post-treatment pain scores, track pain trends across sessions, and assess long-term outcomes. Participants will continue receiving routine care, and therapy will be adjusted based on individual responses.

ELIGIBILITY:
Inclusion Criteria:

* Able to verbalize pain scores
* Oncology patients with acute and/or chronic pain

Exclusion Criteria:

* Patients with Implantable Devices
* Epilepsy
* Pregnancy
* A history of myocardial infarction or ischemic heart disease within the past six months
* History of severe heart arrhythmia or equivalent heart disease
* Open Wounds or Infections at site of electrode placement
* A history of intolerance to transcutaneous electronic nerve stimulation

Ages: 5 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported pain intensity as assessed by the Numerical Rating Scale or the Wong-Baker Faces Pain Scale | Prior to first therapy session and immediately following last therapy session
  The primary outcome is the change in self-reported pain intensity from baseline (prior to the first Scrambler Therapy session) to the post-final Scrambler Therapy session as measured by Numerical Rating Scale (NRS) or Wong-Baker Faces Pain Scale. The patients will rate pain using one of these scales at the beginning and the end of each treatment session with the primary comparison between the pre-first treatment session and the post-final treatment session. Total score range from 0-10, for both scales with a higher score indicating more pain.

SECONDARY OUTCOMES:
Change in pain intensity as assessed by the Numerical Rating Scale or the Wong-Baker Faces Pain Scale. | immediately prior to and immediately following each session
  Intra-session to session change in pain intensity across the full course of a single Scrambler Therapy session. Total score range from 0-10, with a higher score indicating more pain
Change in pain characteristics measured via the PainDETECT questionnaire, comparing responses from first and final sessions. | Prior to first therapy session and immediately after final therapy session
  Total score range from 0-38. A higher score indicates a greater likelihood of neuropathic pain.
Change in number of medications used, daily morphine equivalents for opioids | Prior to first therapy session up to 1 week following last therapy session.
  This will be obtained through medical records.
Change in total dose reduction for neuropathic pain | Prior to first therapy session up to 1 week following last therapy session.
  This will be obtained through medical records.
Durability of pain relief as assessed by the Numerical Rating Scale or the Wong-Baker Faces Pain Scale. | 1 month post therapy sessions, 6 months post therapy sessions
  Total score range from 0-10, with a higher score indicating more pain

CONTACTS AND LOCATIONS:
Overall Officials: Joann Hunsberger, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Children's Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No